CLINICAL TRIAL: NCT06160609
Title: A Phase I/II, Randomized, Open-label Platform Study Utilizing a Master Protocol to Study Belantamab Mafodotin (GSK2857916) as Monotherapy and in Combination With Anti-Cancer Treatments in Participants With Relapsed/Refractory Multiple Myeloma (RRMM)-DREAMM5. Sub-study 1 - Belantamab Mafodotin and aOX40 (GSK3174998) in Combination
Brief Title: Platform Sub-study of Belantamab Mafodotin (GSK2857916) in Combination With aOX40 (GSK3174998) in Participants With RRMM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208887 Sub Study 1; 2019-001138-32 (EudraCT Number)
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belantamab mafodotin + GSK3174998 (Experimental)
  Interventions: Drug: Belantamab Mafodotin; Drug: GSK3174998

INTERVENTIONS:
Drug: Belantamab Mafodotin — Belantamab Mafodotin will be administered.
  Other Names: GSK2857916
Drug: GSK3174998 — GSK3174998 will be administered.
  Other Names: aOX40

SUMMARY:
The primary purpose is to determine the safety and tolerability of belantamab mafodotin in combination with other anti-cancer treatments (in each sub-study), and to establish the recommended Phase 2 dose for each combination treatment to explore in the cohort expansion phase. This study is the sub study of the Master protocol (NCT04126200).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age inclusive or older, at the time of signing the informed consent.
* Participants must have histologically or cytologically confirmed diagnosis of Multiple Myeloma (MM), as defined by the IMWG.
* Participants having at least 3 prior lines of prior anti-myeloma treatments including an immunomodulating agent (IMID) a proteasome inhibitor (PI) and an anti-CD38 monoclonal antibody.
* Participants with a history of autologous stem cell transplant are eligible for study participation when, transplant was >100 days prior to study enrolment and with no active infection(s).
* Participants with Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, unless ECOG less than equal to (<=)2 is due solely to skeletal complications and/or skeletal pain due to MM.
* Participants with measurable disease defined as at least one of the following: Serum M-protein greater than equal to (>=)0.5 gram per deciliter (>=5 gram per liter) or Urine M-protein >=200 milligrams (mg) per 24 hours or Serum free light chain (FLC) assay: Involved FLC level >=10 mg per deciliter (>=100 mg per Liter) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants who have tested positive for Hepatitis B core antibody (HBcAb) can be enrolled if the following criteria are met: Serology result HBcAb+, Hepatitis B surface antigen (HBsAg)-; HBV deoxyribonucleic acid (DNA) undetectable during screening.
* Participants who are currently receiving physiological doses oral steroids (<10 mg/day), inhaled steroids or ophthalmological steroids.

Exclusion Criteria:

* Participants with current corneal epithelial disease except mild punctate keratopathy.
* Participants with evidence of cardiovascular risk.
* Participants with known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to belantamab mafodotin or any of the components of the study treatment. History of severe hypersensitivity to other mAb.
* Participants with active infection requiring antibiotic, antiviral, or antifungal treatment.
* Participants with other monoclonal antibodies within 30 days or systemic anti-myeloma therapy within <14 days.
* Participants with prior radiotherapy within 2 weeks of start of study therapy.
* Participants with prior allogeneic transplant are prohibited.
* Participants who have received prior Chimeric Antigen T cell therapy (CAR-T) therapy with lymphodepletion with chemotherapy within 3 months of screening.
* Participants with any major surgery (other than bone-stabilizing surgery) within the last 30 days.
* Participants with prior treatment with an investigational agent within 14 days or 5 half-lives of receiving the first dose of study drugs, whichever is shorter.
* Participants with >=grade 3 toxicity considered related to prior check-point inhibitors and that led to treatment discontinuation.
* Participants who have received transfusion of blood products within 2 weeks before the first dose of study drug.
* Participants must not receive live attenuated vaccines within 30 days prior to first dose of study treatment or whilst receiving belantamab mafodotin +- partner agent in any sub-study arm of the platform trial and for at least 70 days following last study treatment.
* Participants with presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM.
* Participants with known human immunodeficiency virus (HIV) infection, unless the participant can meet all criteria: a) established anti-retroviral therapy for at least 4 weeks and HIV viral load<400 copies/milliliter (mL) b) cluster of differentiation 4 plus (CD4+) T-cell (CD4+) counts >= 350 cells/microliter (µL) c) No history of Acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the last 12 months in which case the participant would be eligible for CE Phase only.
* Participants with autoimmune disease (current or history) or syndrome that required systemic treatment within the past 2 years.
* Exclusion for a recent (within the past 6 months) history of symptomatic pericarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Fitzroy, Victoria, Australia
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a sub-study of the master study NCT04126200. This sub study was terminated due to lack of efficacy. The study was planned to include two phases - Dose Escalation (DE) and Cohort Expansion (CE) and no participants were enrolled in CE phase as study was early terminated.
Groups:
- 1.9 mg/kg Belantamab Mafodotin + 8mg OX40: Participants with Relapsed/Refractory Multiple Myeloma (RRMM) received 1.9 milligram (mg)/kilogram (kg) belantamab mafodotin intravenous (IV) infusion as powder for solution once every 3 weeks (Q3W) infused over 30- 60 minutes on day 1 of 21-day cycles in combination with 8 mg OX40 IV solution 1 hour after belantamab mafodotin end of infusion (EOI) on day 1 of 21-day cycles.
- 2.5 mg/kg Belantamab Mafodotin + 8mg OX40: Participants with RRMM received 2.5 mg/kg belantamab mafodotin IV infusion as powder for solution Q3W infused over 30- 60 minutes on day 1 of 21-day cycles in combination with 8 mg OX40 IV solution 1 hour after belantamab mafodotin EOI on day 1 of 21-day cycles.
Period: Overall Study
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Started | 6 | 3
Completed (Participants who completed follow-up or who died were considered to have completed the study.) | 6 (1 participant completed the follow-up and 5 participants died) | 3 (1 participant completed the follow-up and 2 participants died)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1.9 mg/kg Belantamab Mafodotin + 8mg OX40: Participants with RRMM received 1.9 milligram (mg)/kilogram (kg) belantamab mafodotin intravenous (IV) infusion as powder for solution once every 3 weeks (Q3W) infused over 30- 60 minutes on day 1 of 21-day cycles in combination with 8 mg OX40 IV solution 1 hour after belantamab mafodotin end of infusion (EOI) on day 1 of 21-day cycles.
- Total: Total of all reporting groups
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40 | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (11.15) | 73.3 (2.31) | 70.4 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: DE Phase: Number of Participants With Dose Limiting Toxicities (DLT)
Description: Criteria for dose-limiting toxicity (DLT) included hematologic indicators such as Grade 3-5 febrile neutropenia and thrombocytopenia with bleeding. Non-hematologic criteria, excluding corneal toxicity, comprise Grade 3-5 toxicities, with exceptions for manageable nausea, vomiting, or diarrhea, controlled Grade 3 hypertension, and events linked to disease progression. Tumor lysis syndrome (TLS) of Grade 3 or 4, successfully managed within 7 days without end-organ damage, is considered. Corneal toxicity, assessed by the GSK corneal grading scale at Grade 4, is a DLT. Other organ-specific toxicities, notably liver toxicity meeting GSK stopping criteria, also qualify as DLTs.
Time Frame: Up to 21 days
Population: DLT Evaluable Population included participants in DE phase who received the first course of treatment containing both agents within a sub-study and followed up within cycle 1 (Each cycle is of 21 days) or withdrew within cycle 1 due to an AE meeting the definition of a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

2. Primary Outcome: DE Phase: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
Participants | 6 | 3

3. Primary Outcome: DE Phase: Number of Participants With Worst-Case Hematology Results by Maximum Grade Increase Post - Baseline Relative to Baseline
Description: Blood samples were collected for the analysis of following hematology parameters: eosinophils, anemia, hemoglobin increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, leukocytosis and white blood cell decreased. The laboratory parameters were graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5. Grade 1 (G1): mild; Grade 2 (G2): moderate; Grade 3 (G3: severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Any worst-case post baseline increase to G1, G2 and G3 are presented.
Time Frame: Baseline (Day 1) and up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
Participants
  Eosinophils, Increase to G1 | 0 | 0
  Eosinophils, Increase to G2 | 0 | 0
  Eosinophils, Increase to G3 | 0 | 0
  Anemia, Increase to G1 | 0 | 2
  Anemia, Increase to G2 | 2 | 0
  Anemia, Increase to G3 | 1 | 0
  Hemoglobin Increased, Increase to G1 | 0 | 0
  Hemoglobin Increased, Increase to G2 | 1 | 0
  Hemoglobin Increased, Increase to G3 | 0 | 0
  Lymphocyte Count Decreased, Increase to G1 | 1 | 2
  Lymphocyte Count Decreased, Increase to G2 | 1 | 0
  Lymphocyte Count Decreased, Increase to G3 | 1 | 0
  Lymphocyte Count Increased, Increase to G1 | 0 | 0
  Lymphocyte Count Increased, Increase to G2 | 0 | 0
  Lymphocyte Count Increased, Increase to G3 | 0 | 0
  Neutrophil Count Decreased, Increase to G1 | 0 | 0
  Neutrophil Count Decreased, Increase to G2 | 2 | 0
  Neutrophil Count Decreased, Increase to G3 | 0 | 0
  Platelet Count Decreased, Increase to G1 | 2 | 2
  Platelet Count Decreased, Increase to G2 | 2 | 0
  Platelet Count Decreased, Increase to G3 | 2 | 0
  Leukocytosis, Increase to G1 | 0 | 0
  Leukocytosis, Increase to G2 | 0 | 0
  Leukocytosis, Increase to G3 | 0 | 0
  White Blood Cell Decreased, Increase to G1 | 1 | 0
  White Blood Cell Decreased, Increase to G2 | 3 | 0
  White Blood Cell Decreased, Increase to G3 | 0 | 0

4. Primary Outcome: DE Phase: Number of Participants With Worst-Case Chemistry Results by Maximum Grade Increase Post - Baseline Relative to Baseline
Description: Blood samples were collected for the analysis of following chemistry parameters: Hypoglycemia, hypoalbuminemia, alkaline phosphatase (ALP) increased, alanine aminotransferase (ALT) increased, aspartate aminotransferase (AST) increased, blood bilirubin increased, creatine kinase (CPK) increased, creatinine increased, gamma glutamyl transferase (GGT) increased, hyperkalemia, blood lactate dehydrogenase (LDH) increased, hypermagnesemia, hypomagnesemia, hypernatremia, hypercalcemia, hypocalcemia and Serum OR Plasma Glomerular Filtration Rate (GFR) from creatinine adjusted for body surface area (BSA) SA (mL/sec/1.73m^2)/chronic kidney disease. The laboratory parameters were graded according to CTCAE version 5. G1: mild; G2: moderate; G3: severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Any worst-case post baseline increase to G1, G2 and G3 are presented.
Time Frame: Baseline (Day 1) and up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
Participants
  Hypoglycemia, Increase to G1 | 0 | 0
  Hypoglycemia, Increase to G2 | 0 | 0
  Hypoglycemia, Increase to G3 | 0 | 1
  Hypoalbuminemia, Increase to G1 | 1 | 0
  Hypoalbuminemia, Increase to G2 | 2 | 0
  Hypoalbuminemia, Increase to G3 | 1 | 0
  ALP Increased, Increase to G1 | 4 | 0
  ALP Increased, Increase to G2 | 0 | 1
  ALP Increased, Increase to G3 | 0 | 0
  ALT Increased, Increase to G1 | 1 | 1
  ALT Increased, Increase to G2 | 0 | 0
  ALT Increased, Increase to G3 | 0 | 0
  AST Increase, Increase to G1 | 4 | 1
  AST Increase, Increase to G2 | 0 | 1
  AST Increase, Increase to G3 | 0 | 0
  Blood bilirubin Increased, Increase to G1 | 0 | 0
  Blood bilirubin Increased, Increase to G2 | 0 | 0
  Blood bilirubin Increased, Increase to G3 | 0 | 0
  CPK Increased, Increase to G1 | 2 | 1
  CPK Increased, Increase to G2 | 0 | 1
  CPK Increased, Increase to G3 | 0 | 0
  Creatinine Increased, Increase to G1 | 3 | 0
  Creatinine Increased, Increase to G2 | 1 | 1
  Creatinine Increased, Increase to G3 | 0 | 0
  GGT Increased, Increase to G1 | 3 | 1
  GGT Increased, Increase to G2 | 1 | 1
  GGT Increased, Increase to G3 | 0 | 0
  Hyperkalemia, Increase to G1 | 1 | 1
  Hyperkalemia, Increase to G2 | 0 | 0
  Hyperkalemia, Increase to G3 | 0 | 0
  LDH increased, Increase to G1 | 2 | 2
  LDH increased, Increase to G2 | 0 | 0
  LDH increased, Increase to G3 | 0 | 0
  Hypermagnesemia, Increase to G1 | 0 | 1
  Hypermagnesemia, Increase to G2 | 0 | 0
  Hypermagnesemia, Increase to G3 | 1 | 0
  Hypomagnesemia, Increase to G1 | 1 | 1
  Hypomagnesemia, Increase to G2 | 0 | 0
  Hypomagnesemia, Increase to G3 | 1 | 0
  Hypernatremia, Increase to G1 | 0 | 0
  Hypernatremia, Increase to G2 | 0 | 0
  Hypernatremia, Increase to G3 | 0 | 0
  Hypercalcemia, Increase to G1 | 1 | 1
  Hypercalcemia, Increase to G2 | 1 | 0
  Hypercalcemia, Increase to G3 | 0 | 0
  Hypocalcemia, Increase to G1 | 0 | 0
  Hypocalcemia, Increase to G2 | 0 | 0
  Hypocalcemia, Increase to G3 | 0 | 0
  GFR from creatinine/Chronic Kidney Disease, Increase to G1 | 0 | 0
  GFR from creatinine/Chronic Kidney Disease, Increase to G2 | 1 | 0
  GFR from creatinine/Chronic Kidney Disease, Increase to G3 | 1 | 0

5. Primary Outcome: Cohort Expansion (CE) Phase: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was defined as the percentage of participants with a confirmed PR or better as the best overall response (i.e., Partial Response [PR], Very Good Partial Response [VGPR], Complete Response [CR], and stringent Complete Response [sCR]), as assessed by the investigator per international myeloma working group (IMWG) (2016). CR defined as negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR defined as CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR defined as serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR defined as ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Up to 170 weeks
Population: Intent to Treat (ITT) population included all the enrolled participants. No participants were enrolled in CE Phase as study got terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: DE Phase: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed partial response (PR) or better (i.e., PR, very good partial response [VGPR], complete response [CR] and stringent complete response [sCR]), according to the International Myeloma Working Group (IMWG) Response Criteria. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
Percentage of participants | 0 | 0

7. Secondary Outcome: CE Phase: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate was defined as the percentage of participants with a confirmed minimal response (MR) or better according to the IMWG Response Criteria. MR is >= 25% but < 49% reduction of serum M-protein and reduction in 24-hour urinary M-protein by 50-89%.
Time Frame: Up to 170 weeks
Population: as for outcome 5
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: DE Phase: Percentage of Participants Achieving Stringent Complete Response (SCR), Complete Response (CR), Very Good Partial Response (VGPR) and Partial Response (PR)
Description: Partial Response [PR], Very Good Partial Response [VGPR], Complete Response [CR], and stringent Complete Response [sCR] as assessed by the investigator per IMWG (2016). CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
Percentage of participants
  Stringent Complete Response (sCR) | 0 | 0
  Complete response (CR) | 0 | 0
  Very Good Partial Response (VGPR) | 0 | 0
  Partial response (PR) | 0 | 0

9. Secondary Outcome: CE Phase: Percentage of Participants Achieving SCR, CR, VGPR and PR
Description: as for outcome 8
Time Frame: Up to 170 weeks
Population: as for outcome 5
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: DE Phase: Plasma Concentrations of Belantamab Mafodotin Antibody-Drug Conjugate (ADC)
Description: Blood samples were collected for PK analysis of belantamab mafodotin Antibody-Drug Conjugate (ADC).
Time Frame: Up to Day 1 (End of Infusion) of Cycle 6 (Each Cycle consist of 21 days)
Population: Pharmacokinetic population included all participants in the safety population from whom at least one PK sample has been obtained and analysed.
Measure: Median (Full Range); unit: nanogram/ millilitre (ng/mL)
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
nanogram/ millilitre (ng/mL)
  Cycle 1 Day 1, Pre-Dose: number analyzed (Participants) | 4 | 3
  Cycle 1 Day 1, Pre-Dose | 0.0 [0 to 0] | 0.0 [0 to 0]
  Cycle 1 Day 1, End Of Infusion | 30100.0 [25900 to 36400] | 43400.0 [31400 to 50000]
  Cycle 1 Day 1, 2 hours | 29450.0 [25100 to 32100] | 39700.0 [29800 to 45800]
  Cycle 1 Day 1, 24 hours | 18300.0 [13700 to 27800] | 30900.0 [20000 to 31000]
  Cycle 1 Day 4 | 9925.0 [6240 to 15500] | 10700.0 [9420 to 15500]
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 8 | 3880.0 [3530 to 4880] | 7180.0 [5170 to 8220]
  Cycle 1 Day 22: number analyzed (Participants) | 1 | 1
  Cycle 1 Day 22 | 1060.0 | 3130.0
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 4 | 3
  Cycle 2 Day 1, Pre-Dose | 1415.0 [878 to 1700] | 1390.0 [679 to 2720]
  Cycle 2 Day 1, End Of Infusion: number analyzed (Participants) | 5 | 3
  Cycle 2 Day 1, End Of Infusion | 27700.0 [24100 to 33000] | 42900.0 [32500 to 54000]
  Cycle 4 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 1
  Cycle 4 Day 1, Pre-Dose | 2635.0 [2190 to 3080] | 2190.0
  Cycle 4 Day 1, End Of Infusion: number analyzed (Participants) | 2 | 1
  Cycle 4 Day 1, End Of Infusion | 28200.0 [27200 to 29200] | 29900.0
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 1 | 1
  Cycle 6 Day 1, Pre-Dose | 3600.0 | 2800.0
  Cycle 6 Day 1, End Of Infusion: number analyzed (Participants) | 1 | 1
  Cycle 6 Day 1, End Of Infusion | 32100.0 | 27500.0

11. Secondary Outcome: CE Phase: Plasma Concentrations of Belantamab Mafodotin Antibody-Drug Conjugate (ADC)
Description: Blood samples were collected for PK analysis of Belantamab Mafodotin Antibody-Drug Conjugate (ADC).
Time Frame: Up to Day 1 (End of Infusion) of Cycle 6 (Each Cycle consist of 21 days)
Population: No participants were enrolled in CE Phase as study got terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: DE Phase: Plasma Concentration of Belantamab Mafodotin Total Antibody
Description: Blood samples were collected for PK analysis of Belantamab mafodotin total antibody.
Time Frame: Up to Day 1 (End of Infusion) of Cycle 6 (Each Cycle consist of 21 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: ng/mL
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
ng/mL
  Cycle 1 Day 1, Pre-Dose: number analyzed (Participants) | 3 | 2
  Cycle 1 Day 1, Pre-Dose | 0.0 [0 to 0] | 0.0 [0 to 0]
  Cycle 1 Day 1, End Of Infusion | 32650.0 [29600 to 36400] | 49500.0 [38200 to 56800]
  Cycle 1 Day 1, 2 hours | 34500.0 [30000 to 37000] | 46000.0 [37800 to 53000]
  Cycle 1 Day 1, 24 hours | 23650.0 [18500 to 32900] | 36700.0 [26600 to 41000]
  Cycle 1 Day 4 | 15900.0 [9950 to 22000] | 21500.0 [16300 to 25100]
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 8 | 9770.0 [7460 to 10400] | 18300.0 [10600 to 21500]
  Cycle 1 Day 22: number analyzed (Participants) | 1 | 0
  Cycle 1 Day 22 | 2620.0 |
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 4 | 3
  Cycle 2 Day 1, Pre-Dose | 4105.0 [2600 to 5170] | 3740.0 [3070 to 8680]
  Cycle 2 Day 1, End Of Infusion: number analyzed (Participants) | 5 | 3
  Cycle 2 Day 1, End Of Infusion | 34000.0 [29300 to 41800] | 52000.0 [40800 to 56200]
  Cycle 4 Day 1, Pre-Dose: number analyzed (Participants) | 3 | 1
  Cycle 4 Day 1, Pre-Dose | 6910.0 [4560 to 11800] | 5430.0
  Cycle 4 Day 1, End Of Infusion: number analyzed (Participants) | 3 | 1
  Cycle 4 Day 1, End Of Infusion | 40500.0 [39100 to 40900] | 33200.0
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 1 | 1
  Cycle 6 Day 1, Pre-Dose | 13100.0 | 8720.0
  Cycle 6 Day 1, End Of Infusion: number analyzed (Participants) | 1 | 1
  Cycle 6 Day 1, End Of Infusion | 47500.0 | 40400.0

13. Secondary Outcome: CE Phase: Plasma Concentration of Belantamab Mafodotin Plasma Total Antibody
Description: Blood samples were collected for PK analysis of Belantamab mafodotin plasma total antibody.
Time Frame: Up to Day 1 (End of Infusion) of Cycle 6 (Each Cycle consist of 21 days)
Population: Pharmacokinetic population included all participants in the safety population from whom at least one PK sample has been obtained and analysed. No participants were enrolled in CE Phase as study got terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: DE Phase: Plasma Concentrations of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis of belantamab mafodotin cys- monomethyl auristatin-F (cys-mcMMAF).
Time Frame: Up to Day 1 (End of Infusion) of Cycle 6 (Each Cycle consist of 21 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: ng/mL
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
ng/mL
  Cycle 1 Day 1, Pre-Dose | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0]
  Cycle 1 Day 1, End Of Infusion | 404.00 [352.0 to 741.0] | 623.00 [343.0 to 735.0]
  Cycle 1 Day 1, 2 hours | 489.00 [338.0 to 811.0] | 527.00 [515.0 to 832.0]
  Cycle 1 Day 1, 24 hours | 766.50 [449.0 to 1760.0] | 1020.00 [722.0 to 1050.0]
  Cycle 1 Day 4 | 360.50 [288.0 to 752.0] | 492.00 [309.0 to 615.0]
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 8 | 120.00 [107.0 to 235.0] | 234.00 [172.0 to 292.0]
  Cycle 1 Day 22: number analyzed (Participants) | 1 | 1
  Cycle 1 Day 22 | 0.00 | 0.00
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 5 | 3
  Cycle 2 Day 1, Pre-Dose | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0]
  Cycle 2 Day 1, End Of Infusion: number analyzed (Participants) | 5 | 3
  Cycle 2 Day 1, End Of Infusion | 384.00 [262.0 to 676.0] | 625.00 [353.0 to 796.0]
  Cycle 4 Day 1, Pre-Dose: number analyzed (Participants) | 3 | 1
  Cycle 4 Day 1, Pre-Dose | 0.00 [0.0 to 0.0] | 0.00
  Cycle 4 Day 1, End Of Infusion: number analyzed (Participants) | 3 | 1
  Cycle 4 Day 1, End Of Infusion | 548.00 [268.0 to 679.0] | 268.00
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 1 | 1
  Cycle 6 Day 1, Pre-Dose | 0.00 | 0.00
  Cycle 6 Day 1, End Of Infusion: number analyzed (Participants) | 1 | 1
  Cycle 6 Day 1, End Of Infusion | 291.00 | 179.00

15. Secondary Outcome: CE Phase: Plasma Concentrations of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: Blood samples were collected for PK analysis of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Time Frame: Up to Day 1 (End of Infusion) of Cycle 6 (Each Cycle consist of 21 days)
Population: as for outcome 13
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: DE Phase: OX40 Concentration When Administered in Combination With Belantamab Mafodotin
Description: Blood samples were collected for PK analysis of OX40 when administered intravenously in combination with belantamab mafodotin.
Time Frame: Up to Day 1 (End of Infusion) of Cycle 6 (Each Cycle consist of 21 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: ng/mL
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
ng/mL
  Cycle 1 Day 1, Pre-Dose | 0.0 [0 to 0] | 0.0 [0 to 0]
  Cycle 1 Day 1, End Of Infusion | 1199.5 [0 to 1478] | 1759.0 [1746 to 2671]
  Cycle 1 Day 1, 24 hours | 1078.0 [712 to 1305] | 1540.0 [1427 to 1974]
  Cycle 1 Day 1, 2-4 hours | 1576.0 [1137 to 1659] | 1888.0 [1785 to 1889]
  Cycle 1 Day 4 | 576.5 [428 to 770] | 889.0 [751 to 1087]
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 8 | 358.0 [0 to 545] | 737.0 [487 to 874]
  Cycle 1 Day 22: number analyzed (Participants) | 1 | 1
  Cycle 1 Day 22 | 0.0 | 326.0
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 5 | 3
  Cycle 2 Day 1, Pre-Dose | 0.0 [0 to 0] | 0.0 [0 to 0]
  Cycle 4 Day 1, Pre-Dose: number analyzed (Participants) | 3 | 1
  Cycle 4 Day 1, Pre-Dose | 0.0 [0 to 551] | 0.0
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 1 | 1
  Cycle 6 Day 1, Pre-Dose | 0.0 | 346.0

17. Secondary Outcome: CE Phase: OX40 Concentration When Administered in Combination With Belantamab Mafodotin
Description: as for outcome 16
Time Frame: Up to Day 1 (End of Infusion) of Cycle 6 (Each Cycle consist of 21 days)
Population: as for outcome 13
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: DE Phase: Number of Participants With Post-baseline Positive Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples were tested in screening assay, and positive samples were further characterized for antibody titers.
Time Frame: Up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

19. Secondary Outcome: CE Phase: Number of Participants With Post-baseline Positive ADAs Against Belantamab Mafodotin
Description: as for outcome 18
Time Frame: Up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
  No participants were enrolled in CE Phase as study got terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: DE Phase: Number of Participants With Post-baseline Positive ADAs Against OX40
Description: as for outcome 18
Time Frame: Up to 170 weeks
Population: Data was not collected.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: CE Phase: Number of Participants With Post-baseline Positive ADAs Against OX40
Description: as for outcome 18
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: DE Phase: Concentration of ADAs Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples were to be further tested in screening assay, and positive samples were further to be characterized for antibody titers.
Time Frame: Up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy. No participants were found positive for ADAs, hence participants were not analyzed for concentration of ADAs.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: CE Phase: Concentration of ADAs Against Belantamab Mafodotin
Description: as for outcome 22
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: DE Phase: Concentration of ADAs Against OX40 When Administered in Combination With Belantamab Mafodotin
Description: as for outcome 22
Time Frame: Up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
  There were no participants with positive ADA results. Hence participants were not analyzed for the concentration of ADA.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: CE Phase: Concentration of ADAs Against OX40 When Administered in Combination With Belantamab Mafodotin
Description: as for outcome 22
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: DE Phase: Number of Participants With Adverse Events of Special Interest (AESI)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. Adverse Events of Special Interest (whether serious or non serious) were collected.
Time Frame: Up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
Participants | 6 | 3

27. Secondary Outcome: CE Phase: Number of Participants With AESI
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: DE Phase: Number of Participants With Any Corneal Events by Maximum Grade as Per CTCAE Grade
Description: The corneal events were graded according to CTCAE version 5. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Results are presented for number of participants with any corneal events by maximum grade as per CTCAE grade.
Time Frame: Up to 170 weeks
Population: Safety Population included all participants who received at least 1 dose of any component of the combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 6 | 3
Participants
  Grade 1 | 1 | 0
  Grade 2 | 3 | 1
  Grade 3 | 0 | 1

29. Secondary Outcome: CE Phase: Number of Participants With Any Corneal Events by Maximum Grade as Per CTCAE Grade
Description: Corneal Events were examined.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: CE Phase: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization until the earliest date of confirmed progressive disease (PD) per IMWG, or death due to any cause.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: CE Phase: Duration of Response (DoR)
Description: DoR is defined as the time from first documented evidence or PR or better until progressive disease per IMWG or death due to progressive disease among participants who achieve confirmed partial response or better.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: CE Phase: Time to Response (TTR)
Description: TTR is defined as the time between the date of randomization and the first documented evidence of response (PR or better), among participants who achieve a response (confirmed PR or better).
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: CE Phase: Overall Survival (OS)
Description: OS is defined as the time from randomization until death due to any cause.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: CE Phase: Number of Participants With AEs and SAEs
Description: AEs and SAEs were collected.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: CE Phase: Number of Participants With AEs Leading to Discontinuation
Description: Number of participants with AEs leading to discontinuation were evaluated.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: CE Phase: Number of Participants With Dose Reduction or Delay
Description: Number of participants with dose reduction or delay were evaluated.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: CE Phase: Number of Participants With Clinically Significant Changes in Hematology Lab Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: eosinophils, anemia, hemoglobin increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, leukocytosis and white blood cell decreased. The laboratory parameters were graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5. Grade 1 (G1): mild; Grade 2 (G2): moderate; Grade 3 (G3: severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: CE Phase: Number of Participants With Clinically Significant Changes in Clinical Chemistry Lab Parameters
Description: Blood samples were collected for the analysis of following chemistry parameters: Hypoglycemia, hypoalbuminemia, alkaline phosphatase (ALP) increased, alanine aminotransferase (ALT) increased, aspartate aminotransferase (AST) increased, blood bilirubin increased, creatine kinase (CPK) increased, creatinine increased, gamma glutamyl transferase (GGT) increased, hyperkalemia, blood lactate dehydrogenase (LDH) increased, hypermagnesemia, hypomagnesemia, hypernatremia, hypercalcemia, hypocalcemia and chronic kidney disease. The laboratory parameters were graded according to CTCAE version 5. G1: mild; G2: moderate; G3: severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade.
Time Frame: Up to 170 weeks
Population: as for outcome 19
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected maximum up to 170 weeks.
Description: Safety set included all participants who received at least one dose of any component of the combination therapy in the combination arm.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40
All-Cause Mortality (participants affected / at risk) | 5/6 | 2/3
Serious Adverse Events (participants affected / at risk) | 6/6 | 1/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 (N=6) | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40 (N=3)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.9 mg/kg Belantamab Mafodotin + 8mg OX40 (N=6) | 2.5 mg/kg Belantamab Mafodotin + 8mg OX40 (N=3)
Keratopathy (Eye disorders) | 2 (2) | 2 (7)
Dry eye (Eye disorders) | 1 (1) | 1 (2)
Vision blurred (Eye disorders) | 1 (2) | 1 (3)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (2) | 0 (0)
Exophthalmos (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Mass (General disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT06160609/Prot_002.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT06160609/SAP_001.pdf